CLINICAL TRIAL: NCT06748586
Title: The Effect of Hyperbaric Oxygen Therapy (HBOT) on Circulating Hematopoietic Stem Cell Population , a Prospective Study.
Brief Title: The Effect of Hyperbaric Oxygen Therapy on Circulating Hematopoietic Stem Cell Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0165-24
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Circulating Hematopoietic Stem Cells
Keywords: hyperbaric oxygen therapy
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: hyperbaric oxygen therapy (2ATA, 100% oxygen)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperbaric oxygen therapy (HBOT) active treatment (Active Comparator): The HBOT protocol is 90 minutes, 5 times/week, for at least 40 sessions, 100% oxygen at 2 ATA with five-minute air breaks every 20 minutes
  Interventions: Device: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — The HBOT protocol is 90 minutes, 5 times/week, for at least 40 sessions, 100% oxygen at 2 ATA with five-minute air breaks every 20 minutes. Investigational product: Multiplace hyperbaric oxygen chamber (Haux Starmed 2700, Germany) located at the Sagol center for hyperbaric medicine and research, Shamir (Assaf-Harofeh) Medical Center, Israel.

SUMMARY:
Hematopoietic stem cells (HSCs), which govern the production of all blood lineages, transition through a series of functional states characterized by expansion during fetal development, functional quiescence in adulthood, and decline upon aging.

Although research on aging has for a long time been relatively descriptive, much progress has been made in the past decade to uncover the molecular drivers of biological aging. One such drivers relates to stem cell exhaustion.

The amount and the function of HSCs decline in humans along aging. This decline is characterized by different changes such as signaling, epigenetic, cell surface markers etc. Various studies have been conducted to identify HSCs surface markers using flow cytometry.

Exposure to HBOT induce stem cells proliferation mobilization of stem progenitor cells (SPCs) in both animal and humans studies, and the number of SPCs remain elevated in blood over the course of 20 HBOT .

Additionally, Heyboer et al have found dose response curve between the HBOT protocol and circulating CD34+ and CD45-dim (stem cells potential markers): increasing the treatment pressure from 2.0 ATA to 2.5 ATA increased the concentration of circulating stem cells.

The aim of the current study is to evaluate the effect of HBOT on circulating hematopoietic stem cells, in the peripheral blood of patients who are candidate for HBOT.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients aged 20-80 who are intendent to start HBOT for other indication that are willing to give blood samples for measurements of circulating stem cells.

Exclusion Criteria:

1. Active or recent infection within the last month
2. Active malignancy.
3. History of hematopoietic disease
4. Low B12 or iron levels
5. Inability to sign the informed consent form
6. Leucocytes ˂4000 or ˃10,000

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
hematopoietic stem cells evaluation | Change from Baseline immediately after the intervention
  Blood test will be withdrawn for hematopoietic stem cells evaluation, CBC and chemistry. Evaluation of the hematopoietic stem cells population in PBMCs in different HBOT time points. Hematopoietic Stem cells will be identified by Flow cytometry immunostaining with the following markers: CD34, CD38- , CD45, CD45RA and CD90. A negative control will be an unstained tube and a tube containing CD45+CD34+ and CD38+, a positive control will be the Isotope control for each marker. The tube including the CD38- marker will be specific for the stem cells population.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sagol Center for Hyperbaric Medicine and Research Shamir Medical Center (Assaf Harofeh), Zrifin, Israel, Israel

IPD SHARING:
Plan to Share IPD: Undecided